CLINICAL TRIAL: NCT03257475
Title: Evaluation of Vaginal Dose in Cervical Cancer Patients Treated With Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Liu Zi, Professor, Xi'an Jiaotong University
Other Study IDs: XIAN J
Record Dates: First submitted 2017-08-14; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cervical Cancer
Keywords: cervical cance; vaginal radiation injury; PIBS; R-V; VRL
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Brachytherapy — Intracavitary irradiation starts at the end of the external beam radiation using image-guided CT/SIM.CT/SIM (transverse axis) is done to complete 3/2D treatment planning. Measurement VRL, PIBS and PIBS ± 2cm, R-V were recorded; Brachytherapy plan: Point A: 24-30Gy/4-5f, or 21-28Gy/3-4f HR-CTV: ≥85Gy, IR-CTV 65Gy dose records

SUMMARY:
Cervical cancer is the most common malignant in women with the average five-year overall survival rate as high as 70%. Radiation therapy is the main treatment for cervical cancer. Vagina is one of the important organ at risk and also a target organ in the treatment of cervical cancer patients. Vaginal radiation has serious related complications that affect the quality of life of patients and therefore needs much clinical attention. But due to lack of sufficient evidence, the clinical dose to the vagina is limited. ICRU-89 defined the recto-vaginal reference point (R-V) as a reference point for vaginal dose assessment. However, the R-V position is affected by applicator placement, vaginal packing and other factors hence the dose point only do not represent the entire vaginal radiation dose resulting in some clinical limitations. The latest research in Europe proposed that PIBS(Posterior-Inferior Border of Symphysis) / PIBS ± 2cm and VRL (vaginal reference length) may be more reasonable to use to assess vagina radiation doses, but it remains to be further clinically investigated. Therefore, this study intends to perform radical radiotherapy in cervical cancer patients and also by recruiting local and foreign hospitals into this study by recording its PIBS/ PIBS ± 2cm, VRL, R-V point dose, acute and chronic radiation injury incidence of vagina and other useful data. T-test and chi-square will be used to compare the data between Asian and European women. Correlation analysis will be used to determine if there is a relation between R-V and PIBS point dose. Furthermore, logic and or COX regression model to evaluate PIBS / PIBS ± 2cm and R-V point doses of vaginal radiation injury relationships, while exploring other relevant factors causing vaginal radiation injury. This is eventually expected to provide a scientific, simple and reliable reference point for vaginal dose assessment and clinical dose limit.

DETAILED DESCRIPTION:
1. a detailed record of the irradiation dose and R-V point dose for all patients PIBS / PIBS ± 2cm, VRL data were taken.
2. according to CTCAE v3.0 standard, accurate and detailed record of patient treatment, after treatment of 2 years and the incidence of vaginal complications were recorded.
3. COX regression model was used to find dose-effect relationship between the reference point and vaginal complications.

Clinical Scheme:

Inclusion criteria: Pathologically confirmed cervical cancer patients, FIGO stage ⅠA- ⅣA patients who underwent radical radiotherapy, Any pathological type

Exclusion criteria: FIGO staging of cervical cancer ⅢA; Age > 60 years due to vaginal stenosis during the treatment course

1. pre-treatment: Abdominal and Chest CT scan before treatment. Patients were given pelvic MRI after EBRT to measure VRL before the start of brachytherapy.
2. 3DCRT / IMRT was used and according to RTOG target outlined recommendation dose of 46-50Gy / 23-25f; recording PIBS WP and R-V WP dose.
3. Intracavitary irradiation starts at the end of the external beam radiation using image-guided CT / SIM. catheterization of full bladder. Patients were advice to have empty rectum before CT scan

   The first treatment method:
   1. Catheterization: placement of catheter inside bladder and injection of contrast agent-containing 7ml liquid
   2. Place uterine and vaginal applicator device (must double the bulb), vaginal orifices ball from 3cm, and record
   3. Vaginal packing with gauze is done to keep the applicator fixed.
   4. Barium into the rectum and anal canal.
   5. CT/SIM (transverse axis) is done to complete 3D / 2D treatment planning. measurement VRL, PIBS and PIBS ± 2cm, R-V were recorded;
   6. Brachytherapy plan: Point A: 24-30Gy / 4-5f, or 21-28Gy / 3-4f HR-CTV: ≥85Gy, IR-CTV 65Gy dose records;
4. Concurrent chemotherapy: DDP 30-40mg / m2 * 5w or T 135mg / m2D1 + DDP 30mg / m2 d1-3;
5. vaginal washing method is every day from the beginning of radiation therapy for six months. After 6 months, it was done twice per week for 2 years.
6. vaginal radiation complications were recorded according to CTCAE 3.0 standard
7. Gynecological examination and MRI was performed before radiotherapy and brachytherapy treatment and also after the entire treatment period. Patients follow-up was done on the 1,3,6,9,12,18 and 24th month after treatment during which vaginal radiation complication were evaluated according to CTCAE 3.0 standard
8. COX regression model was used to find dose-effect relationship between the reference point and vaginal complications.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed cervical cancer patients;
* FIGO stage ⅠA- ⅣA patients who underwent radical radiotherapy;
* Any pathological type

Exclusion Criteria:

* FIGO staging of cervical cancer ⅢA;
* Age > 60 years

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pathologically confirmed cervical cancer patients, FIGO stage ⅠA-ⅣA patients who underwent radical radiotherapy except ⅢA, Any pathological type.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
PIBS/PIBS±2cm dose in Gy | two weeks
  record the PIBS/PIBS±2cm dose by planning system
VRL in centimeter | two weeks
  measure the VRL in MRI
R-V dose in Gy | two weeks
acute and chronic radiation injury incidence of vagina | two years
  acute and chronic radiation injury incidence of vaginaas assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Juan Wang, Ph.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fidarova EF, Berger D, Schussler S, Dimopoulos J, Kirisits C, Georg P, Bachtiary B, Potter R. Dose volume parameter D2cc does not correlate with vaginal side effects in individual patients with cervical cancer treated within a defined treatment protocol with very high brachytherapy doses. Radiother Oncol. 2010 Oct;97(1):76-9. doi: 10.1016/j.radonc.2010.05.005. Epub 2010 Jun 17. PMID 20561694
- [Background] Rai B, Dhanireddy B, Patel FD, Kumari R, Oinam AS, Simha V, Sharma S. Vaginal dose, toxicity and sexual outcomes in patients of cervical cancer undergoing image based brachytherapy. Asian Pac J Cancer Prev. 2014;15(8):3619-23. doi: 10.7314/apjcp.2014.15.8.3619. PMID 24870767
- [Background] Murakami N, Kasamatsu T, Sumi M, Yoshimura R, Harada K, Kitaguchi M, Sekii S, Takahashi K, Yoshio K, Inaba K, Morota M, Ito Y, Itami J. Vaginal tolerance of CT based image-guided high-dose rate interstitial brachytherapy for gynecological malignancies. Radiat Oncol. 2014 Jan 23;9:31. doi: 10.1186/1748-717X-9-31. PMID 24456669
- [Background] Prescribing, Recording, and Reporting Brachytherapy for Cancer of the Cervix. J ICRU. 2013 Apr;13(1-2):NP. doi: 10.1093/jicru/ndw027. No abstract available. PMID 27335496
- [Background] Kirchheiner K, Nout RA, Lindegaard JC, Haie-Meder C, Mahantshetty U, Segedin B, Jurgenliemk-Schulz IM, Hoskin PJ, Rai B, Dorr W, Kirisits C, Bentzen SM, Potter R, Tanderup K; EMBRACE Collaborative Group. Dose-effect relationship and risk factors for vaginal stenosis after definitive radio(chemo)therapy with image-guided brachytherapy for locally advanced cervical cancer in the EMBRACE study. Radiother Oncol. 2016 Jan;118(1):160-6. doi: 10.1016/j.radonc.2015.12.025. Epub 2016 Jan 9. PMID 26780997
- [Background] Susko M, Craciunescu O, Meltsner S, Yang Y, Steffey B, Cai J, Chino J. Vaginal Dose Is Associated With Toxicity in Image Guided Tandem Ring or Ovoid-Based Brachytherapy. Int J Radiat Oncol Biol Phys. 2016 Apr 1;94(5):1099-105. doi: 10.1016/j.ijrobp.2015.12.360. Epub 2015 Dec 19. PMID 26883564
- [Background] Westerveld H, de Leeuw A, Kirchheiner K, Dankulchai P, Oosterveld B, Oinam A, Hudej R, Swamidas J, Lindegaard J, Tanderup K, Potter R, Kirisits C; EMBRACE Collaborative Group. Multicentre evaluation of a novel vaginal dose reporting method in 153 cervical cancer patients. Radiother Oncol. 2016 Sep;120(3):420-427. doi: 10.1016/j.radonc.2016.05.002. Epub 2016 May 26. PMID 27237058
- [Derived] Wang J, Zhang KS, Wang T, Liu Z, Wang RH, Zhang FQ, Yu L, Ran L, He JL, Wang YL, Wei LC, Shi M, Wang GQ, Wu CQ, Kang QJ, Yang J, Li S, Yang FY, Liu BG, Liu JY, Shi F, Su J, Yuan W, Drokow EK. Vaginal dose of radical radiotherapy for cervical cancer in China: a multicenter study. BMC Cancer. 2019 Dec 16;19(1):1219. doi: 10.1186/s12885-019-6423-5. PMID 31842811